CLINICAL TRIAL: NCT04904354
Title: AcQBlate Force Sensing Ablation System US IDE Study for Atrial Fibrillation (AcQForce AF)
Brief Title: AcQBlate Force Sensing Ablation System US IDE Study for Atrial Fibrillation
Acronym: AcQForce AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company no longer doing clinical studies
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP-16; CLP-16-EU (Other: Acutus Medical, Inc.); NCT04941391 (obsolete NCT alias)
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Two distinct, non-randomized cohorts of subjects will be included; a PAF population and a PerAF population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Paroxysmal atrial fibrillation (Experimental): Subjects schedule for a de novo ablation of paroxysmal atrial fibrillation
  Interventions: Device: AcQBlate® Force Sensing Ablation System
- Persistent atrial fibrillation (Experimental): Subjects schedule for a de novo ablation of persistent atrial fibrillation
  Interventions: Device: AcQBlate® Force Sensing Ablation System

INTERVENTIONS:
Device: AcQBlate® Force Sensing Ablation System — Catheter ablation of accessible pulmonary veins with the endpoint of creating electrical isolation for each targeted vein. Additional left and right atrial targets may be ablated as clinically indicated.

SUMMARY:
The AcQForce AF clinical study is a prospective, multi-center, non-randomized global clinical study.

DETAILED DESCRIPTION:
The AcQForce AF clinical study is a prospective, multi-center, non-randomized global clinical study designed to demonstrate the safety and efficacy of the AcQBlate Force Sensing System in the ablation treatment of symptomatic, drug-refractory atrial fibrillation in two subject cohorts: paroxysmal atrial fibrillation, and persistent atrial fibrillation. Data will be used to support pre-market approval applications (PMAs).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 to 80 years at time of consent
2. Clinically indicated and scheduled for a de novo catheter ablation of symptomatic PAF or PerAF.
3. Refractory to Antiarrhythmic Drug (AAD) treatment
4. Willing and able to provide written informed consent to participate in the study and agree to comply with all follow-up visits and evaluations for the duration of the study.

Exclusion Criteria:

1. In the opinion of the investigator, any contraindication to the planned atrial ablation, including anticoagulation contraindications or sepsis.
2. Continuous episodes of AF Duration:

   1. PAF: AF duration lasting longer than 7 days
   2. Persistent AF: AF duration lasting longer than 12-months.
3. Atrial arrhythmias secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause.
4. An implantable cardiac defibrillator (ICD) or pacemaker.
5. Previous history of left atrial ablation (including surgical treatment) for AF/AT/AFL.
6. Structural heart disease or cardiac history as described below:

   1. Left ventricular ejection fraction (LVEF) < 40% based on transthoracic echocardiogram (TTE) within the previous 180-days.
   2. Left atrial size > 55 mm based on transthoracic echocardiogram (TTE) measurement of the anteroposterior diameter, parasternal long-axis view in M Mode and performed within the previous 180-days.
   3. Evidence of heart failure (NYHA Class III or IV)
   4. Previous cardiac surgery, ventriculotomy, or atriotomy (excluding atriotomy for coronary artery bypass).
   5. Previous cardiac valvular surgical or percutaneous procedure, or prosthetic valve.
   6. Coronary artery bypass graft (CABG) within the last 180-days or coronary angioplasty (PTCA) procedure within the last 90-days.
   7. Unstable angina or ongoing myocardial ischemia.
   8. Myocardial infarction within the previous 180-days (sub-endocardial infarct within previous 90-days).
   9. Severe uncontrolled systemic hypertension (systolic pressure > 240 mm Hg, diastolic pressure > 140 mm Hg) recorded within the last 30 days.
   10. Moderate or severe valvular heart disease (stenosis or regurgitation).
   11. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder.
   12. Presence of a left atrial appendage occlusion device.
   13. Previous PV stenting or evidence of PV stenosis.
7. Presence of Left Atrial Thrombus
8. Body Mass Index (BMI) > 42 kg/m2
9. Estimated Glomerular Filtration Rate (eGFR) of <40 mL/min/1.73 m2 (by Modification of Diet in Renal Disease formula)
10. History of blood clotting or bleeding disease.
11. ANY prior history of documented cerebral infarct, or systemic embolism (excluding post-operative deep vein thrombosis (DVT)).
12. History of chronic obstructive pulmonary disease (COPD) requiring oral or IV steroid use in the previous 12-months.
13. History of obstructive sleep apnea not currently being treated.
14. Pregnant or lactating (current or anticipated during study follow-up).
15. Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements for this study.
16. Any other condition that, in the judgment of the Investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, terminal illness with a life expectancy of less than two years, extensive travel away from the research center).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjects who are free from device and/or procedure related Major Adverse Events (MAEs) | 12 months
  Subjects free from a composite list of pre-specified procedure/device related Major Adverse Events (MAEs)
Proportion of subjects demonstrating freedom from AF/AT/AFL following a blanking period | 12 months
  Freedom from recurrence of atrial arrhythmias

SECONDARY OUTCOMES:
Recording of all serious adverse events/device effects | 12 months
  Recording of all serious adverse events/device effects

IPD SHARING:
Plan to Share IPD: No